CLINICAL TRIAL: NCT02835170
Title: Evaluation of Efficacy and Safety of Intramuscular Administration of Autologous Total Immunoglobulin G in Adolescent and Adult Patients With Moderate-to-severe Atopic Dermatitis: A Randomized, Double-blind, Placebo-controlled Study
Brief Title: Study of Autologous Total Immunoglobulin G Therapy for Atopic Dermatitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Dong-Ho Nahm, Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AJIRB-MED-SMP-13-359
Record Dates: First submitted 2016-06-08; First posted 2016-07-15 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Dermatitis, Atopic
Keywords: Immunoglobulin G; Treatment
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous immunoglobulin (Experimental): Intramuscular injection of autologous immunoglobulin (IgG)
  Interventions: Biological: Autologous immunoglobulin
- Placebo (Placebo Comparator): Intramuscular injection of normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Autologous immunoglobulin — Autologous immunoglobulin (total IgG) aseptically purified from the autologous plasma will be administered to the patients by intramuscular injection, once a week for 7 weeks (total 8 injections).
  Other Names: AIGT
  Arms: Autologous immunoglobulin
Other: Placebo — Saline will be administered to the patients by intramuscular injection, once a week for 7weeks (total 8 injections).
  (In addition, autologous immunoglobulin is colorless and odorless, injection volume is same between autologous immunoglobulin and saline)
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled parallel group study on the efficacy and safety of intramuscular injections of autologous immunoglobulin in patients with moderate-to-severe atopic dermatitis.

DETAILED DESCRIPTION:
Children and adult patients with moderate-to-severe atopic dermatitis (age ≥ 13 years) whose clinical conditions have not been effectively controlled by current standard medical therapies (topical moisturizers, topical corticosteroids, topical calcineurin inhibitors, and oral antihistamines) for more than 2 months will be include.

This is a randomized, double-blind, placebo-controlled parallel group study on the efficacy and safety of intramuscular injections of autologous immunoglobulin in patients with moderate-to-severe atopic dermatitis. After providing informed consent, patients will be assessed for study eligibility at the baseline visit. Patients will undergo screening within 28 days prior to randomization as "wash out period", and during the screening period, treatment with medications (including systemic corticosteroids and systemic immunomodulating agents) for atopic dermatitis will be wash-out for at least 28 days prior to baseline (exclude moisturizers).

At screening, plasma will be separated from patients' venous blood (400ml) aseptically and autologous immunoglobulin (total IgG) will be purified from the plasma by chromatography using Protein A during the screening period. Patients will be randomized in a 1:1 ratio to receive weekly treatment with autologous immunoglobulin or placebo (normal saline) will be administrated by intramuscular injection, once a week for 7 weeks (total 8 injections).

The investigators will evaluate the clinical efficacy and safety of intramuscular injections of autologous immunoglobulin in those patients with moderate-to-severe atopic dermatitis by measuring changes in the standardized clinical severity scoring system for atopic dermatitis (SCORAD) values, Eczema Area and Severity index (EASI) and quality of life together with laboratory parameters in blood samples before and after treatment. Systemic corticosteroids as a rescue treatment will be prescribed to control unacceptable symptoms of atopic dermatitis at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Suitability of autologous blood donation criteria
2. Current standard medical therapies more than 2 months and moderate-to-severe atopic dermatitis
3. ≥10% lesion body surface area (BSA) of atopic dermatitis involvement in area

Exclusion Criteria:

1. Patients under the age of 13 year.
2. Patients who are unable to agree on their own (emergency patients, patients with mental disability, patients with limited capacity to consent due to stroke or delirium caused by diabetes).
3. Patients with severe disease whose expected survival duration is less than 3 months.
4. Pregnancy or planned pregnancy within 1 year
5. Skin condition not appropriate for blood sampling and transfusion
6. The standardized clinical severity scoring system for atopic dermatitis (SCORAD) values <25 (Mild atopic dermatitis)

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-04-02 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

PRIMARY OUTCOMES:
Change in EASI index | baseline to week 16
  The Eczema Area and Severity index (EASI) is a used in clinical practice and clinical trials to evaluates the clinical severity of atopic dermatitis

SECONDARY OUTCOMES:
EASI-50 | baseline to week 16
  Achieving reduction in the EASI score greater than index from baseline
Change in SCORAD values | baseline to week 16
  Standardized clinical severity scoring system for atopic dermatitis (SCORAD) value is a used in clinical practice and clinical trials to evaluates the clinical severity of atopic dermatitis
Change in BSA | baseline to week 16
  percentage change in body surface area
Change in DLQI index | baseline to week 16
  Dermatologic assessment tools that patients to test the reliability and validity 10-item Dermatology Life Quality Index (DLQI) questionnaire in patients with atopic dermatitis

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Ho Nahm, M.D., Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou university hosiptal, Suwon, Gyeong-gi Do, South Korea

IPD SHARING:
Plan to Share IPD: Yes